CLINICAL TRIAL: NCT01863550
Title: Randomized Phase III Trial of Bortezomib, Lenalidomide, and Dexamethasone (VRd) Versus Carfilzomib, Lenalidomide, and Dexamethasone (CRd) Followed by Limited or Indefinite Duration Lenalidomide Maintenance in Patients With Newly Diagnosed Symptomatic Multiple Myeloma (ENDURANCE)
Brief Title: Bortezomib or Carfilzomib With Lenalidomide and Dexamethasone in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1A11; NCI-2012-02608 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E1A11; E1A11; s17-00040; E1A11 (Other: ECOG-ACRIN Cancer Research Group); E1A11 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2013-05-06; First posted 2013-05-29 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; carfilzomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (bortezomib, lenalidomide, dexamethasone) (Experimental): Patients receive bortezomib SC or IV on days 1, 4, 8, and 11 of courses 1-8 and days 1 and 8 of courses 9-12; lenalidomide PO daily on days 1-14; and dexamethasone PO daily on days 1, 2, 4, 5, 8, 9, 11, and 12 of courses 1-8 and days 1, 2, 8, and 9 of courses 9-12. Treatment repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Quality-of-Life Assessment
- Arm B (carfilzomib, lenalidomide, dexamethasone) (Experimental): Patients receive carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16; lenalidomide PO daily on days 1-21; and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 4 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Quality-of-Life Assessment
- Arm C (lenalidomide) (Experimental): Patients receive lenalidomide PO daily on days 1-21. Treatment repeats every 4 weeks for 24 courses in the absences of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Quality-of-Life Assessment
- Arm D (lenalidomide) (Experimental): Patients receive lenalidomide PO daily on days 1-21. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Bortezomib — Given SC or IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
  Arms: Arm A (bortezomib, lenalidomide, dexamethasone)
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
  Arms: Arm B (carfilzomib, lenalidomide, dexamethasone)
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
  Arms: Arm A (bortezomib, lenalidomide, dexamethasone); Arm B (carfilzomib, lenalidomide, dexamethasone)
Other: Laboratory Biomarker Analysis — Optional correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies bortezomib, lenalidomide, and dexamethasone to see how well they work compared to carfilzomib, lenalidomide, and dexamethasone in treating patients with newly diagnosed multiple myeloma. Bortezomib and carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Lenalidomide may help the immune system kill abnormal blood cells or cancer cells. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether bortezomib, lenalidomide, and dexamethasone are more or less effective than carfilzomib, lenalidomide, and dexamethasone in treating patients with multiple myeloma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall survival between two strategies of lenalidomide maintenance following induction with a proteasome inhibitor? immunomodulatory drug (IMiD) combination: limited duration of maintenance (24 months) versus indefinite maintenance therapy until disease progression.

II. To compare progression-free survival between bortezomib, lenalidomide, and dexamethasone (VRd) and carfilzomib, lenalidomide, and dexamethasone (CRd) induction followed by lenalidomide maintenance in patients with newly diagnosed symptomatic multiple myeloma.

SECONDARY OBJECTIVES:

I. To compare the progression-free survival between two strategies of lenalidomide maintenance following induction with a proteasome inhibitor?IMiD combination: limited duration of maintenance (24 months) or indefinite maintenance therapy until disease progression.

II. To compare induction rates of response between VRd and CRd arms. III. To evaluate time to progression, duration of response and overall survival between VRd and CRd induction therapy.

IV. To compare induction rates of toxicity between VRd and CRd arms. V. To evaluate toxicity during lenalidomide maintenance. VI. To compare minimal residual disease (MRD) negative rates between VRd and CRd arms at end of induction therapy.

TERTIARY OBJECTIVES:

I. To compare the short and long-term health-related quality of life impact between the two strategies of lenalidomide maintenance.

II. To compare the impact on health-related quality of life between VRd and CRd induction therapy.

III. To evaluate the association between early induction response and change in health-related quality of life.

IV. To describe changes in health-related quality of life during the induction, active maintenance and observation phases.

V. To evaluate correlation between treatment adherence during maintenance and health-related quality of life.

VI. To compare MRD negative rates between the two strategies of lenalidomide maintenance.

VII. To compare MRD negative rates between VRd and CRd arms during induction therapy.

VIII. To examine patterns of change in MRD levels over time and examine conversion from detectable to MRD negative status.

IX. To evaluate agreement and association between International Myeloma Working Group (IMWG) and MRD based disease-free status.

X. To describe the mutational profile of newly diagnosed multiple myeloma. XI. To identify mutations associated with resistance to VRd and CRd induction therapy.

XI. To identify expression profiles associated with MRD negative status with each induction therapy.

XII. To determine the ability of MRD status at induction end to predict short-term and long-term overall and progression-free survival.

XIII. To determine the effects of tobacco, operationalized as combustible tobacco (1a), other forms of tobacco (1b), and environmental tobacco exposure (ETS) (1c) on provider-reported cancer-treatment toxicity (adverse events [both clinical and hematologic] and dose modifications).

XIV. To determine the effects of tobacco on patient-reported physical symptoms and psychological symptoms.

XV. To examine quitting behaviors and behavioral counseling/support and cessation medication utilization.

XVI. To explore the effect of tobacco use and exposure on treatment duration, relative dose intensity, and therapeutic benefit.

OUTLINE:

INDUCTION: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive bortezomib subcutaneously (SC) or intravenously (IV) on days 1, 4, 8, and 11 of courses 1-8 and days 1 and 8 of courses 9-12; lenalidomide orally (PO) daily on days 1-14; and dexamethasone PO daily on days 1, 2, 4, 5, 8, 9, 11, and 12 of courses 1-8 and days 1, 2, 8, and 9 of courses 9-12. Treatment repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16; lenalidomide PO daily on days 1-21; and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 4 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: After completion of induction therapy (or completion of at least 6 courses in Arm A but stopped early due to unacceptable toxicity, or at least 4 courses in Arm B but stopped early due to unacceptable toxicity), patients are then randomized to 1 of 2 maintenance treatment arms.

ARM C: Patients receive lenalidomide PO daily on days 1-21. Treatment repeats every 4 weeks for 24 courses in the absences of disease progression or unacceptable toxicity.

ARM D: Patients receive lenalidomide PO daily on days 1-21. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP I: Patients must be diagnosed with symptomatic standard-risk multiple myeloma (SR-MM) as defined by all of the following (except gene expression profile [GEP]70 status if unknown):

  * No evidence of t(14;16) by fluorescence in situ hybridization (FISH) testing on bone marrow or not available
  * No evidence of t(14:20) by FISH testing on bone marrow or not available
  * No evidence of deletion 17p by FISH testing on bone marrow
  * FISH should be from within 90 days of registration

    * NOTE: If the FISH result states that no immunoglobulin heavy chain (IgH) abnormality is present, both t(14;16) and t(14;20) can be considered negative; in addition, if the patient has a t(11;14) or t(4;14) translocation present, they can be considered negative for t(14;16) and t(14;20); if testing for t(14;16) or t(14;20) could not be performed for lack of sufficient material or non-availability of the probe in the test panel, patients can be enrolled on the study
  * Standard Risk GEP70 signature within the past 90 days (only if GEP has been done and results are available)

    * NOTE: GEP testing is NOT a requirement for the study; if the test has been done, patients found to have a GEP70 status of high-risk will not be eligible
  * Serum lactate dehydrogenase (LDH) =< 2 x upper limit of normal (ULN) within the past 28 days
  * No more than 20% circulating plasma cells on peripheral blood smear differential or 2,000 plasma cells/microliter on white blood cell (WBC) differential of peripheral blood within the past 90 days

    * NOTE: This is NOT the plasma cell % from the marrow aspirate
* STEP I: Patients must have measurable or evaluable disease as defined by having one or more of the following, obtained within 28 days prior to randomization:

  * >= 1 g/dL monoclonal protein (M-protein) on serum protein electrophoresis
  * >= 200 mg/24 hours (hrs) of monoclonal protein on a 24 hour urine protein electrophoresis
  * Involved free light chain >= 10 mg/dL or >= 100 mg/L AND abnormal serum immunoglobulin kappa to lambda free light chain ratio (< 0.26 or > 1.65)
  * Monoclonal bone marrow plasmacytosis >= 30% (evaluable disease)
  * Serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP), and serum free light chain (FLC) assay are required to be performed within 28 days prior to randomization; a bone marrow biopsy and/or aspirate is required within 28 days if bone marrow is being followed for response

    * NOTE: UPEP (on a 24-hour collection) is required, no substitute method is acceptable; urine must be followed monthly if the baseline urine M-spike is >= 200 mg/24 hr; please note that if both serum and urine M-components are present, both must be followed in order to evaluate response
    * NOTE: The serum free light chain test is required to be done if the patient does not have measurable disease in the serum or urine; measurable disease in the serum is defined as having a serum M-spike >= 1 g/dL; measurable disease in the urine is defined as having a urine M-spike >= 200 mg/24 hr
* STEP I: Hemoglobin >= 8 g/dL (obtained within 28 days prior to randomization)
* STEP I: Untransfused platelet count >= 75,000 cells/mm^3 (obtained within 28 days prior to randomization)
* STEP I: Absolute neutrophil count >= 1000 cells/mm^3 (obtained within 28 days prior to randomization)
* STEP I: Calculated creatinine clearance >= 30 mL/min (obtained within 28 days prior to randomization)
* STEP I: Bilirubin =< 1.5 mg/dL (obtained within 28 days prior to randomization)
* STEP I: Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) and serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) < 2.5 times the upper limit of normal (obtained within 28 days prior to randomization)
* STEP I: Patients must have received no more than one cycle (4 weeks or less) of prior chemotherapy and no more than 160 mg of prior dexamethasone (or equivalent dose of prednisone) for treatment of symptomatic myeloma; they should not have been exposed to lenalidomide, bortezomib or carfilzomib for treatment of symptomatic myeloma; prior radiation therapy to symptomatic lesions is allowed provided there are no residual toxicity related to radiation and blood counts that meet the study requirements
* STEP I: Prior systemic glucocorticoid use for the treatment of non-malignant disorders is permitted; prior or concurrent topical or localized glucocorticoid therapy to treat non-malignant comorbid disorders is permitted
* STEP I: Patients must not have active, uncontrolled seizure disorder; patients must have had no seizures in the last 6 months
* STEP I: Patients must not have uncontrolled intercurrent illness including uncontrolled hypertension, symptomatic congestive heart failure, unstable angina, uncontrolled cardiac arrhythmia, uncontrolled psychiatric illness or social situation that would limit compliance with the study, or a prior history of Stevens Johnson syndrome
* STEP I: Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 (performance status [PS] 3 allowed if secondary to pain)
* STEP I: Patients with monoclonal gammopathy of undetermined significance or asymptomatic multiple myeloma are not eligible
* STEP I: Patients must not have grade 2 or higher peripheral neuropathy by Common Terminology Criteria for Adverse Events (CTCAE) 4.0
* STEP I: Patients must not have active, uncontrolled infection
* STEP I: Patients may have a history of current or previous deep vein thrombosis or pulmonary embolism but must be willing to take some form of anti-coagulation as prophylaxis if they are not currently on full-dose anticoagulation
* STEP I: Patients should not have New York Heart Association classification III or IV heart failure or myocardial infarction within the previous 6 months
* STEP I: Patients with a history of prior malignancy are eligible provided they were treated with curative intent and do not require active therapy (currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma ?in situ? of the cervix or breast are not excluded)
* STEP I: Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide throughout the entire duration of study treatment, and for 28 days after the last dose of lenalidomide; FCBP must also agree to ongoing pregnancy testing; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure; female subjects must agree to use contraception or abstinence for 30 days after last dose of carfilzomib

  * A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months
* STEP I: Sexually active males must be willing to use a condom (even if they have undergone a prior vasectomy) while having intercourse, while taking lenalidomide and for 28 days after stopping lenalidomide; male subjects must also agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation from lenalidomide; male subjects must be willing to use condoms for 90 days after discontinuation of carfilzomib
* STEP I: The following patients will be excluded:

  * Pregnant women
  * Nursing women
* STEP I: Human immunodeficiency virus (HIV) infection is not excluded; known HIV positive patients must meet the following criteria:

  * Cluster of differentiation (CD)4 cell count >= 350/mm^3
  * No history of acquired immune deficiency syndrome (AIDS)-related illness
  * Not currently prescribed zidovudine or stavudine
* STEP I: Patient enrolling to this study must agree to register to the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist
* STEP II: Patients must have complete induction without experiencing progression or patients must have received at least 6 cycles on Arm A and 4 cycles on Arm B but stopped induction therapy due to adverse events
* STEP II: Step 2 registration must be within 6 weeks of completing step 1 therapy
* STEP II: Patients must not have received any non-protocol therapy outside of the assigned induction therapy including stem cell transplant
* STEP II: ECOG performance status 0, 1, or 2 (PS 3 allowed if secondary to pain)
* STEP II: Any adverse event related to step 1 therapy must have resolved to grade 2 or less
* STEP II: Hemoglobin >= 8 g/dL (within 28 days prior to randomization to Step II)
* STEP II: Platelet count >= 75,000 cells/mm^3 (within 28 days prior to randomization to Step II)
* STEP II: Absolute neutrophil count >= 1000 cells/mm^3 (within 28 days prior to randomization to Step II)
* STEP II: Calculated creatinine clearance >= 30 mL/min (within 28 days prior to randomization to Step II)
* STEP II: Bilirubin =< 1.5 mg/dL (within 28 days prior to randomization to Step II)
* STEP II: SGPT (ALT) and SGOT (AST) < 2.5 times the upper limit of normal (within 28 days prior to randomization to Step II)
* STEP II: Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide throughout the entire duration of study treatment, and for 28 days after the last dose of lenalidomide; FCBP must also agree to ongoing pregnancy testing; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure

  * A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months
* STEP II: Sexually active males must be willing to use a condom (even if they have undergone a prior vasectomy) while having intercourse, while taking lenalidomide and for 28 days after stopping lenalidomide; male subjects must also agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation from lenalidomide; males must agree to use contraception and agree to not donate sperm for at least 90 days after the last day of carfilzomib
* STEP II: The following patients will be excluded:

  * Pregnant women
  * Nursing women
* STEP II: Patient enrolling to this study must agree to register to the mandatory RevAssist program and be willing and able to comply with the requirements of RevAssist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1087 (Actual)
Dates: Start 2013-12-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2034-02-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) for the maintenance analysis | From the maintenance randomization to death due to any cause or, censored at the date last known alive, assessed up to 15 years
  The Kaplan-Meier (KM) method will be used to describe the overall survival function by arm. Sensitivity analysis will be done to evaluate OS in the subset of eligible patients and censoring patients at time of non-protocol therapy.
Progression-free survival for the induction analysis | From the induction randomization until the earlier of progression or death due to any cause, assessed up to 15 years
  The Kaplan-Meier method will be used to describe the progression-free survival function by arm using all data while ignoring maintenance.

SECONDARY OUTCOMES:
Progression-free survival for the maintenance analysis | From the maintenance randomization until the earlier of progression or death due to any cause, assessed up to 15 years
  Weighted Cox regression will be used.
Overall survival for the induction analysis | From induction randomization to death due to any cause, or censored at the date last known alive, assessed up to 15 years
  The KM method will be used.
Response rates including partial response (PR), very good partial response (VGPR), immunofixation negative complete response (IF-CR) and complete response (CR) | At 2.8 months
  Will be compared between induction arms using Fisher?s exact test.
Response rates including PR, VGPR, IF-CR and CR | At 8.3 months
  Will be compared between induction arms using Fisher?s exact test.
Time to progression (TTP) for the induction analysis | From the induction randomization to progression, or censored at the date of last disease evaluation for those without progression reported, assessed up to 15 years
  TTP distributions will be estimated by induction arm using Kaplan-Meier methods.
Duration of response (DOR) for the induction analysis | From first objective response (partial response or better) since induction randomization until the earlier of progression or death due to any cause, or censored at date of last disease evaluation for those without events reported, assessed up to 15 years
  Duration of response will be estimated using Kaplan-Meier methods in the subset of patients achieving partial response or better while on induction therapy.
Incidence of overall grade 3 or higher non-hematologic toxicity and grade 3 or higher toxicity by type during induction, active maintenance and observation phases using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 15 years
  Fisher?s exact test will be used.
Incidence of grade 2 or higher peripheral neuropathy and cardiac toxicity during induction phase assessed using CTCAE version 5.0 | Up to 36 weeks
  Fisher?s exact test will be used.
Minimal residual disease (MRD) negative rates | At 8.3 months after induction randomization
  MRD evaluation by multiparametric flow cytometry will be conducted and patients classified as MRD negative, MRD positive or not evaluable. At each time point, MRD negative rates with two-sided 95% exact confidence intervals on each arm will be estimated. Patterns of change over time in MRD will also be evaluated using longitudinal regression analysis with general linear mixed effects models and GEE semi-parametric models. MRD negative rates will be compared between either induction or maintenance arms depending on the assessment time point using the Mantel-Haenszel test stratified either on intent to transplant at progression or induction arm (Step 1 and 2 stratification factors, respectively).
Change in the Functional Assessment of Cancer Therapy-Neurotoxicity Trial Outcome Index (FACT-Ntx TOI) for the transition to maintenance analysis | From week 36 (the end) of induction therapy to week 24 (end of course 6) of maintenance therapy
  Will be analyzed using linear mixed models.
Change in the FACT-Ntx TOI for the short-term maintenance analysis | From the end of 2 years of maintenance to 3 years post maintenance randomization
  Will be analyzed using linear mixed models.
Change in the FACT-Ntx TOI for the long-term maintenance analysis | From the end of 2 years of maintenance to 5 years post maintenance randomization
  Will be analyzed using linear mixed models.
Change in the FACT-Ntx TOI for the end of induction analysis | From baseline (induction randomization) to 36 weeks (end) of induction therapy
  Will be analyzed using linear mixed models.
Change in the FACT-Ntx TOI for the early induction analysis | From baseline (induction randomization) to 2.8 months of induction therapy
  Will be analyzed using linear mixed models.
Levels and changes in the FACT-Ntx TOI and Functional Assessment of Cancer Therapy- Multiple Myeloma (FACT-MM) during induction, active maintenance and observation phases | Up to 15 years
  Will be analyzed using linear mixed models.
Time to worsening of FACT-Ntx TOI for the induction analysis | From the baseline assessment at induction randomization to a decrease of 7 points, assessed up to 15 years
  Will be analyzed with KM methods and Cox regression.
Time to worsening of FACT-MM for the maintenance analysis | From the baseline assessment at maintenance randomization to a decrease of 4 points, assessed up to 15 years
  Will be analyzed with KM methods and Cox regression.

OTHER OUTCOMES:
MRD negative rates | At 2.8 months after induction randomization
  MRD evaluation by multiparametric flow cytometry will be conducted and patients classified as MRD negative, MRD positive or not evaluable. At each time point, MRD negative rates with two-sided 95% exact confidence intervals on each arm will be estimated. Patterns of change over time in MRD will also be evaluated using longitudinal regression analysis with general linear mixed effects models and GEE semi-parametric models. MRD negative rates will be compared between either induction or maintenance arms depending on the assessment time point using the Mantel-Haenszel test stratified either on intent to transplant at progression or induction arm (Step 1 and 2 stratification factors, respectively).
MRD negative rates | At 2 years after maintenance randomization
  MRD evaluation by multiparametric flow cytometry will be conducted and patients classified as MRD negative, MRD positive or not evaluable. At each time point, MRD negative rates with two-sided 95% exact confidence intervals on each arm will be estimated. Patterns of change over time in MRD will also be evaluated using longitudinal regression analysis with general linear mixed effects models and GEE semi-parametric models. MRD negative rates will be compared between either induction or maintenance arms depending on the assessment time point using the Mantel-Haenszel test stratified either on intent to transplant at progression or induction arm (Step 1 and 2 stratification factors, respectively).
MRD negative rates | At 3 years after maintenance randomization
  MRD evaluation by multiparametric flow cytometry will be conducted and patients classified as MRD negative, MRD positive or not evaluable. At each time point, MRD negative rates with two-sided 95% exact confidence intervals on each arm will be estimated. Patterns of change over time in MRD will also be evaluated using longitudinal regression analysis with general linear mixed effects models and GEE semi-parametric models. MRD negative rates will be compared between either induction or maintenance arms depending on the assessment time point using the Mantel-Haenszel test stratified either on intent to transplant at progression or induction arm (Step 1 and 2 stratification factors, respectively).
Change in mutation status | Baseline up to 15 years
  Descriptive statistics (absolute frequencies, percentages, mean, standard deviation [SD], median, range) will be used to characterize the study cohort by mutation incidence and expression levels at all time-points.
Change in gene expression levels | Baseline up to 15 years
  Descriptive statistics (absolute frequencies, percentages, mean, SD, median, range) will be used to characterize the study cohort by mutation incidence and expression levels at all time-points. Association of genotype data (binary) with categorical baseline patient and disease characteristics will be evaluated using chi-squared test or, if appropriate, Cochran-Armitage trend test. The Wilcoxon-rank sum test or, if appropriate, the Jonckheere-Terpstra test for trend will be used to assess differential expression levels with baseline patient and disease characteristic groups. The Kaplan-Meier method will be used to estimate progression-free and overall survival distributions and Cox regression to estimate hazard ratios by genotype status.
Circulating plasma cells and plasma cell proliferation | Up to 15 years
  With samples submitted pre-registration, multiparametric flow cytometry will quantify circulating plasma cells (cPC) in terms of number of clonal events/150,000 collected total events and plasma cell proliferation in terms of the plasma cell labeling index (PCLI) percentage. The Kaplan-Meier method will be used to estimate induction progression-free survival and overall survival distributions and Cox regression used to estimate hazard ratios by dichotomized cPC and PCLI.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (920):
- United States (909):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Veteran's Administration Medical Center, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Yale-New Haven Shoreline Medical Center, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Presence Saint Joseph Hospital-Chicago, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - AMITA Health Cancer Institute and Outpatient Center, Hinsdale, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health Bloomington, Bloomington, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc - Jefferson Boulevard, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - The Community Hospital, Munster, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Mary Bird Cancer Center/Saint Tammany Parish, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center/Terrebonne General Medical Center, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - York Hospital, York Village, Maine
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute?Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Huron Valley-Sinai Hospital, Commerce, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Assarian Cancer Center, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Saint Joseph Health System-Tawas City, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Bhadresh Nayak MD PC-Warren, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Nevada Cancer Specialists-Saint Rose, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - Nevada Cancer Specialists?Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - Children's Specialty Center of Nevada II, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Nevada Cancer Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Haywood Infusion Center, Clyde, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Health, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ashland Memorial Medical Center, Ashland, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center - Eau Claire, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Puerto Rico (11):
  - Advance Oncology Center, Aguadilla
  - Doctor's Cancer Center-Arecibo, Arecibo
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Hematologia Oncologia San Pablo, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Primary Care Physician Group, San Juan
  - San Juan City Hospital, San Juan
  - Centro de Hematologia y Oncologia del Sur, Santa Isabel

REFERENCES:
- [Derived] Kumar SK, Jacobus SJ, Cohen AD, Weiss M, Callander N, Singh AK, Parker TL, Menter A, Yang X, Parsons B, Kumar P, Kapoor P, Rosenberg A, Zonder JA, Faber E Jr, Lonial S, Anderson KC, Richardson PG, Orlowski RZ, Wagner LI, Rajkumar SV. Carfilzomib or bortezomib in combination with lenalidomide and dexamethasone for patients with newly diagnosed multiple myeloma without intention for immediate autologous stem-cell transplantation (ENDURANCE): a multicentre, open-label, phase 3, randomised, controlled trial. Lancet Oncol. 2020 Oct;21(10):1317-1330. doi: 10.1016/S1470-2045(20)30452-6. Epub 2020 Aug 28. PMID 32866432